CLINICAL TRIAL: NCT06889064
Title: A Randomized, Open-label, Single Oral Dose, Three-arm, Parallel Design, Phase 1 Study to Evaluate the Pharmacokinetic, Pharmacodynamic Characteristics and the Safety After Administration by Doses of BR1400-1, BR1400-2, BR1400-3 in Healthy Volunteers
Brief Title: A Study to Evaluate the Pharmacokinetic, Pharmacodynamic Characteristics and the Safety After Administration by Doses of BR1400-1, BR1400-2, BR1400-3 in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boryung Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BR-FMS-CT-120
Record Dates: First submitted 2025-03-17; First posted 2025-03-21 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Essential Hypertension
MeSH Terms: conditions — Essential Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- BR1400-1 (Experimental)
  Interventions: Drug: BR1400-1
- BR1400-2 (Experimental)
  Interventions: Drug: BR1400-2
- BR1400-3 (Experimental)
  Interventions: Drug: BR1400-3

INTERVENTIONS:
Drug: BR1400-1 — One tablet administered alone
  Arms: BR1400-1
Drug: BR1400-2 — One tablet administered alone
  Arms: BR1400-2
Drug: BR1400-3 — One tablet administered alone
  Arms: BR1400-3

SUMMARY:
The purpose of this clinical study is to evaluate the pharmacokinetic, pharmacodynamic characteristics and the safety after administration by doses of "BR1400-1", "BR1400-2", "BR1400-3" in healthy volunteers

ELIGIBILITY:
Inclusion Criteria:

* Those who have body mass index (BMI) of 18.0kg/m2 to 30.0kg/m2 at screening visit.

  * For men, Those who weigh 50 kg or more
  * For women, Those who weigh 45 kg or more
* Those who agree to rule out the possibility of their and their spouses' or sexual partners' pregnancy by using methods of contraception accepted in clinical trial* from the date of consent to 7 days after the last administration and disagree to provide their sperm or ovum.

  * Methods of contraception accepted in clinical trial: Combined use of non hormonal intrauterine device, vasectomy, tubal ligation, and barrier methods (male condom, female condom, cervical cap, contraceptive diaphragm, sponge, etc.) or combined use of two or more barrier methods if spermicide is used.
* Those who spontaneously decide to participate and sign written consent to observe the subject's compliance during this clinical trial after listening to and understanding sufficient explanation of the purpose and contents of this clinical trial, characteristics of the Investigational products, expected adverse events, etc.

Exclusion Criteria:

* Those who have taken drugs that induce and inhibit metabolizing enzymes such as barbiturate within 30 days prior to the first day of administration or have taken ethical drugs, over the counter drugs, herbal medicines, health functional foods concerned about affecting this clinical trial within 10 days before the first administration date. (however, participation is possible considering pharmacokinetics and pharmacodynamics such as Interaction of investigational products, half-life of concomitant drugs, etc.)
* Those who have participated in bioequivalence tests or other clinical trials and administered their investigational products within 6 months before the first administration date(However, the termination for participation in other clinical trials are based on the last administration date of their investigational products)
* Those who have a medical history of gastrointestinal diseases (ex. crohn's disease, ulcerative colitis, etc.) or gastrointestinal resection (Except for simple appendectomy, hernia surgery) that may affect the absorption of drugs or have gastrointestinal diseases
* Those who can't discontinue a diet (ex. raw grapefruit, grapefruit juice or food containing grapefruit, etc.) that may affect the absorption, distribution, metabolism, and excretion of the drug within 48 hours before the first administration date
* In the case of a female subject, pregnant woman or those suspected pregnancy or lactating woman.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2024-09-24 (Actual); Primary Completion 2024-10-08 (Actual); Study Completion 2024-10-08 (Actual)

PRIMARY OUTCOMES:
AUCt | 0-48 hours after administration
  Area under the plasma drug concentration-time curve from 0 to time t
Cmax | 0-48 hours after administration
  Maximum concentration of drug in plasma

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul Bumin Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No